CLINICAL TRIAL: NCT00006169
Title: Behavioral Treatment of Weight Gain in CF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Purpose: Prevention
Other Study IDs: Stark (completed); 50092
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Cystic Fibrosis
Keywords: Nutrition; Behavior Therapy; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavioral Treatment

SUMMARY:
The current study examines the efficacy of two treatments to help children with cystic fibrosis (CF) meet their dietary calorie requirements of 120% to 150% of the recommended daily allowance of energy and the effect of these treatments on weight gain and maintenance. One treatment provides children with CF and their parents nutrition education about the best foods for meeting their dietary needs. The second treatment gives children with CF and their families similar nutritional information plus behavioral parenting methods for motivating children to eat the recommended foods. Children with CF and their families are seen weekly for 7 treatment sessions across 9 weeks for the active phase of treatment. Families are then followed for 2 years after treatment in order to better understand how long the treatments are effective and to determine the health benefits of better nutrition status and weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Weight percentile for age or height below 40th for age and sex
* Pancreatic insufficiency

Exclusion Criteria:

* Developmental delays
* Pseudomonas cepacia
* Supplemental enteral or parenteral nutrition

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1996-06; Study Completion 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Lori Stark, Principal Investigator — Children's Hospital & Medical Center
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Children's Hospital Medical Center, Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Derived] Stark LJ, Quittner AL, Powers SW, Opipari-Arrigan L, Bean JA, Duggan C, Stallings VA. Randomized clinical trial of behavioral intervention and nutrition education to improve caloric intake and weight in children with cystic fibrosis. Arch Pediatr Adolesc Med. 2009 Oct;163(10):915-21. doi: 10.1001/archpediatrics.2009.165. PMID 19805710